CLINICAL TRIAL: NCT03106948
Title: Balloon Angioplasty of Dialysis AV Fistulae: Effect of Local Delivery of Inhibitors of Lysyl Oxidase (LysoLox) on Serial Angioplasty and Time to Restenosis
Brief Title: Delivery of Inhibitors of Lysyl Oxidase (LysoLox) on Serial Angioplasty and Time to Restenosis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southeast Renal Research Institute (Other)
Collaborators: Dialysis Clinic, Inc. (Industry)
Responsible Party: Principal Investigator, James A. Tumlin MD, Principal Investigator, Southeast Renal Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Lysyl Oxidase (LysoLox)
Record Dates: First submitted 2017-02-15; First posted 2017-04-11 (Actual); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Arteriovenous Fistula Occlusion
MeSH Terms: interventions — Ascorbic Acid; Penicillamine

STUDY DESIGN:
Intervention Model Description: subjects will be assigned in an open labeled manner to Group 1 (Placebo), Group-2 (Ascorbic Acid), or Group-3 (Ascorbic acid & D-penicillamine). Thus, there will be 10 placebo controls, 10 ascorbic acid patients, and 10 ascorbic acid and D-penicillamine patients. Subjects treated with ascorbic acid in combination with D-penicillamine may have the longest periods between serial angioplasties. Moreover, subjects receiving combination therapy may have greater post-angioplasty luminal diameters.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Low frequency angioplasty (Placebo Comparator): Subjects who have had 0-1 angioplasty during the 12 months prior to randomization. Subjects will have endoluminal biopsy prior to angioplasty but will not have insertion of the ACT drug delivery catheter
  Interventions: Drug: Placebo
- Moderate frequency angioplasty (Active Comparator): Subjects who have had 2-3 angioplasties during the 12 months prior to randomization. Subjects will have endoluminal biopsy prior to angioplasty followed by insertion of the ACT drug delivery catheter where ascorbic acid (10.0 µM) will be injected following conventional balloon angioplasty
  Interventions: Drug: Ascorbic Acid
- High frequency angioplasty (Active Comparator): High frequency angioplasty defined by 4 or more angioplasties 12 months prior to randomization. Subjects will receive ascorbic acid (10.0 µM) in combination with D-penicillamine (25 µM) will be injected following conventional balloon angioplasty
  Interventions: Drug: Cuprimine Oral Product

INTERVENTIONS:
Drug: Placebo — Subject will undergo endoluminal biopsy prior to angioplasty but will NOT undergo insertion of the ACT drug delivery catheter
  Arms: Low frequency angioplasty
Drug: Ascorbic Acid — Subject will undergo endoluminal biopsy prior to angioplasty followed by insertion of the ACT drug delivery catheter where ascorbic acid (10.0 µM) will be injected following conventional balloon angioplasty
  Arms: Moderate frequency angioplasty
Drug: Cuprimine Oral Product — Subject will undergo endoluminal biopsy prior to angioplasty followed by insertion of the ACT drug delivery catheter where ascorbic acid (10.0 µM) in combination with D-penicillamine (25 µM) will be injected following conventional balloon angioplasty
  Other Names: D-Penicillamine
  Arms: High frequency angioplasty

SUMMARY:
The narrowing of Dialysis Fistulae or Grafts is a near universal problem in patients with end-stage renal disease (ESRD) and requires patients to undergo repeated angioplasty or mechanical opening of the fistula.

DETAILED DESCRIPTION:
The failure of dialysis accesses remains a leading cause of morbidity and medical costs among ESRD subjects. The underlying etiology for dialysis access failure is uniformly due to progressive narrowing of the vessel lumen leading to stasis and thrombosis of the access. The luminal narrowing of arteriovenous fistulae (AVFs) is due to progressive hyperplasia of vessel intima and subsequent infiltration of smooth muscle cells into the vessel media. Areas of stenosis within AVFs are characterized by dense neointimal hyperplasia, infiltration of vascular smooth muscle cells and expansion of extracellular matrix material. Additionally, varying types of vascular injury increase the rate of collagen and elastin deposition within the medial and serosal areas of the vessel.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and < 90 years old
* Receiving stable out-subject hemodialysis for a minimum of 3 months
* Have a lower arm or upper arm AVF that has been cleared for use by the vascular surgeon or interventional nephrologist
* Have agreed to participate voluntarily and signed and dated an IRB approved, subject informed consent form
* Dysfunctional Dialysis Fistula: Any subject with

  * Two or more venous pressure readings exceeding 250 mmHg for a minimum of 5 minutes at a blood flow of 500mls/min within a single dialysis run AND a documented reduction in KT/V by > 0.2; OR
  * Patients with venous pressures > 250 mm Hg on two or more days within a 30 day period OR
  * Patients who on physical exam are found to have palpable obstructions, post-stenotic dilation of the access or evidence of prolonged post-dialysis bleeding.
* Any patient with one of the above conditions will be to have a dysfunctional AVF. This definition will be applied to the screening of study subjects as well as the determination of recurrent fistula dysfunction at 12 months.

Exclusion Criteria:

* Scheduled for surgical revision of the fistula;
* Have been in another investigational (non-approved) drug or device study within the previous 30 days;

  **have a known allergy to any component of the investigational product (drug or device)
* Subjects with a "Hero Graft" will be excluded from the study
* Subjects having received a stent for correction of a prior stenosis will be excluded from the trial
* Subjects with more than > 3 hemodynamically significant stenosis at one time (with the exception of a central venous stenosis)
* Subjects who are pregnant will be excluded from the trial (pregnancy test will be performed on subjects of child bearing potential). A urine pregnancy test will be utilized.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-01-31 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Patients treated with ascorbic acid in combination with D-penicillamine will have longer periods between serial angioplasties over 12-month period. Additionally, subjects receiving combination therapy may have greater post-angioplasty luminal diameters. | 12 months
  Subjects are followed for 12 months and monitored for signs of fistula dysfunction. When the patient's fistula becomes dysfunctional they will be referred for a fistulogram. The time between serial fistulograms will be recorded as a secondary endpoint. Patients who are referred for a repeat fistulogram and having a luminal narrowing of greater than 70% will undergo a second intimal biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: James A Tumlin, MD, Principal Investigator — Southeast Renal Research Institute
Locations (1):
- Southeast Renal Research Institute, Chattanooga, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided